CLINICAL TRIAL: NCT02580682
Title: San-fu Herbal Patch and San-fu Moxibustion for Persistent Allergic Rhinitis: a Randomized Controlled Clinical Trial
Brief Title: Sanfu Herbal Patch and Sanfu Moxibustion for Persistent Allergic Rhinitis: a Controlled Clinical Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hubei Provincial Collaborative Innovation Center of Preventive Treatment by Acupuncture and Moxibust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XTCX2014-SFT
Record Dates: First submitted 2015-10-18; First posted 2015-10-20 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2017-04

CONDITIONS: Patch,Chinese Herb; Moxibustion; Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Moxibustion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Since the treatments in this study are visualized, it is not feasible to blind the patients and therapists.Therefore, the outcome assessors will be blinded, they will not participate in the recruitment, study design and the treatment
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sanfu herbal patch (Experimental): one kind of acupoint application which used in hot dog days of summer,The formula of the patch consists of Huang Qi (Astagalus Membranaceus), Fu Zi (Aconiti Lateralis Radix Praeparata), Yan Hu Suo (Rhizoma Corydalis), Xi Xin (Herba asarum), Bai Jie Zi (Semen Sinapis Albae), and Rou Gui (Cortex Cinnamomi) at a ratio of 2:2:1:1:2:1.The bilateral Feishu (BL13), Pishu (BL20), Shenshu (BL23), Neiguan (PC6), and Guanyuan (CV4) acupoints were selected for treatment
  Interventions: Drug: Sanfu herbal patch
- Sanfu moxibustion (Experimental): use moxibustion in hot dog days of summer,and adopting the indirect moxibustion box method at the bilateral BL13, BL20, and BL23 acupoints
  Interventions: Drug: Sanfu moxibustion
- Sanfu herbal patch and Sanfu moxibustion (Experimental): use herbal patch and moxibustion together in hot dog days
  Interventions: Drug: Sanfu herbal patch and moxibustion
- controlled (No Intervention): patients in this group will not accept herbal patch or moxibustion therapy in these 3 years. After the 3-year experimental period they will be offered corresponding treatments for free as well, so they are in our wait list.

INTERVENTIONS:
Drug: Sanfu herbal patch — The formula of the patch consists of Huang Qi (Astagalus Membranaceus), Fu Zi (Aconiti Lateralis Radix Praeparata), Yan Hu Suo (Rhizoma Corydalis), Xi Xin (Herba As5ari), Bai Jie Zi (Semen Sinapis Albae) and Rou Gui(Cortex Cinnamomi), in a proportion of 2:2:1:1:2:1.
  Arms: Sanfu herbal patch
Drug: Sanfu moxibustion — Moxibustion is a kind of thermal therapy without any feeling of pain or swell.Moxibustion exerts its therapeutic effect by thermal power and the application of moxa.
  Arms: Sanfu moxibustion
Drug: Sanfu herbal patch and moxibustion — use Sanfu moxibustion followed by Sanfu herbal patch
  Arms: Sanfu herbal patch and Sanfu moxibustion

SUMMARY:
To observe the efficacy of Sanfu herbal patch and Sanfu moxibustion on persistent allergic rhinitis,and comparing the differences between the combination of these 2 methods with each method alone.

ELIGIBILITY:
Inclusion criteria

Patients recruited to this study must meet the following inclusion criteria:

1. Males or females aged between 5 and 60 years.
2. Each PAR patient must be diagnosed by an otolaryngologist using the following diagnostic criteria: major symptoms of paroxysm rhinocnesmus, continuous sneezing, nasal obstruction, and significant quantities of clear and thin nasal mucus, accompanied by symptoms of hyposmia and itching of the eyes and throat. These symptoms should last for or add up to 1 hour a day. The attacks should occur for more than 4 weeks and at last for at least 4 days each week.
3. One of 2 laboratory results is positive: skin prick test or serum high circulating levels of allergen-specific IgE antibody detected by a specific blood test for allergy called a radioallergosorbent (RAST) test
4. The course of the disease is more than 1 year.
5. Voluntary signing of an informed consent form.
6. No current participation in any other clinical trials. Exclusion criteria

Patients with any of the following conditions will be excluded:

1. Allergies to the herbal medicines, a moxa smoke or adhesive tape applied in this study, and the skin at the specific acupoint has physical scars or breakage.
2. Patients with other allergic diseases, such as allergic asthma.
3. Patients who received acupuncture and moxibustion treatment, Chinese herbal medicine, nasal inhalation of herbal medicine, physical therapy or other external treatment for AR within the last 4 weeks
4. Patients who received immune therapy or systematic hormonotherapy in the past 1 year.
5. Pregnant women, lactating women, or women preparing for pregnancy in 2 years.
6. Patients with serious medical disorders such as congenital heart disease, severe nephropathy, mental diseases, and infectious diseases including tuberculosis, hepatitis, and AIDS.

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Total Nasal Symptom Score(TNSS) | three years
  In TNSS, symptoms of nasal congestion , sneezing, nasal itching and rhinorrhea are assessed by scores ranging from 0 to 3. A score of 0 indicates no symptoms, 1 for mild symptoms that are easily tolerated, 2 for awareness of symptoms which are bothersome but tolerable and 3 is reserved for severe symptoms that are hard to tolerate and interfere with daily activity .TNSS is calculated by adding the score for each symptom together

SECONDARY OUTCOMES:
visual analogue scale (VAS) | three years
  VAS is a 10cm scale to assess the impact of AR on life quality ranging from score of 0 to 10, which stands for "no impact" to "serious impact
Rhinitis Quality of Life Questionnaire (RQLQ) | three years
  The RQLQ contains 28 questions to evaluate impairment of everyday life caused by symptoms of nose and eyes. Seven dimensions will be assessed, including daily life, sleep, non-nosal/optical symptoms, practical problems, nosal symptoms, optical symptoms and emotion. Every question should be answered by scores: 0 - not trouble, 1 - any trouble at all, 2 - somewhat troubled, 3 - moderately troubled, 4 - quite a bit of trouble, 5 - very troubled, 6 - extremely troubled.
36-item Short-Form Health Survey (SF-36) | three years
  SF-36 consists of 36 items categorized as eight dimensions: social functioning (two items), role limitation-emotion (three items), mental health (five items), physical functioning (ten items), role limitation-physical (four items), bodily pain (two items), vitality (four items), general health (five items) and one question of health change in recent one year.

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei university of TCM, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
we have recruited approximately sixty patients in tha last year, informations including contacting numbers, medical history, questionnaires and follow-up materials, we have not decided in which way we could share these data.